CLINICAL TRIAL: NCT03847779
Title: Microcirculatory Vasomotor Function in Response to Acute Exercise in Type 2 Diabetes With Peripheral Neuropathy
Brief Title: Microcirculatory Vasomotor Changes in Type 2 Diabetes With Peripheral Neuropathy
Acronym: NEUROMICRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UAPV-012019-AVJ
Record Dates: First submitted 2019-01-28; First posted 2019-02-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Neuropathy Peripheral; Small Vessel Disease of Diabetes Mellitus; Vasodilation; Vasoconstriction
Keywords: vasomotion
MeSH Terms: conditions — Diabetic Angiopathies; Aneurysm | interventions — RE1-silencing transcription factor; Exercise; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-neuropathy (Experimental): Type 2 diabetic without neuropathy:
  * Negative findings on Semmes-Weinstein monofilament
  * Neuropathy symptom score (NSS) <3
  * Negative findings on Nerve Check and Diabetic Peripheral Neuropathy check.
  Interventions by means of Laser Doppler Flowmetry and Laser Speckle Imaging:
  * "rest" cutaneous microcirculation (perfusion and vasomotion)
  * "Exercise" cutaneous microcirculation (perfusion and vasomotion)
  * "Foot lowering" cutaneous microcirculation (perfusion and vasomotion)
  * "Hyperthermia" cutaneous microcirculation (perfusion and vasomotion)
  * blood sampling
  * heart rate variability at rest
  * pedometer during 4 days
  * international Physical Activity Questionary
  * Qualify of Life questionary (EQVOD)
  Interventions: Other: "Rest"; Other: "Exercise"; Other: "Foot lowering"; Other: "Hyperthermia"
- Neuropathy (Experimental): Type 2 diabetic with neuropathy
  * Positive findings on Semmes-Weinstein monofilament
  * Neuropathy symptom score (NSS) >3
  * Positive findings on Nerve Check and Diabetic Peripheral Neuropathy check.
  Interventions by means of Laser Doppler Flowmetry and Laser Speckle Imaging:
  * "rest" cutaneous microcirculation (perfusion and vasomotion)
  * "Exercise" cutaneous microcirculation (perfusion and vasomotion)
  * "Foot lowering" cutaneous microcirculation (perfusion and vasomotion)
  * "Hyperthermia" cutaneous microcirculation (perfusion and vasomotion)
  * blood sampling
  * heart rate variability at rest
  * pedometer during 4 days
  * international Physical Activity Questionary
  * Qualify of Life questionary (EQVOD)
  Interventions: Other: "Rest"; Other: "Exercise"; Other: "Foot lowering"; Other: "Hyperthermia"
- Controls (Experimental): matched for age, sexe and BMI with diabetic patients.
  Interventions by means of Laser Doppler Flowmetry and Laser Speckle Imaging:
  * "rest" cutaneous microcirculation (perfusion and vasomotion)
  * "Exercise" cutaneous microcirculation (perfusion and vasomotion)
  * "Foot lowering" cutaneous microcirculation (perfusion and vasomotion)
  * "Hyperthermia" cutaneous microcirculation (perfusion and vasomotion)
  * blood sampling
  * heart rate variability at rest
  * international Physical Activity Questionary
  * Qualify of Life questionary (EQVOD)
  Interventions: Other: "Rest"; Other: "Exercise"; Other: "Foot lowering"; Other: "Hyperthermia"

INTERVENTIONS:
Other: "Rest" — Cutaneous perfusion and vasomotion assessment at rest in supoine position
Other: "Exercise" — Cutaneous perfusion and vasomotion assessment after the 6minute-wlaking test
Other: "Foot lowering" — Cutaneous perfusion and vasomotion assessment after foot lowering
Other: "Hyperthermia" — Cutaneous perfusion and vasomotion assessment during hyperthermia

SUMMARY:
Microcirculatory flow is subject to cyclic changes under the influence of heart rate, respiration, myogenic activity, neurogenic factors and endothelial factors. Microcirculatory oscillations (vasomotion) contribute significantly to tissue perfusion. Vasomotion analysis allowed to discriminate normoglycemic subjects, prediabetic subjects and diabetic subjects. Furthermore, changes in vasomotion can precede the emergence of global signs of microangiopathy complications in type 2 diabetes. In fact, few studies reported impaired vasomotion in type 2 diabetes with peripheral neuropathy. Vasomotion analysis after vasodilator (6-min walking test and hyperthermia) and after vasoconstrictor (foot lowering) stimulus could be an effective diagnostic tool to sharpen the diagnostic.

Objectives and Methodology: to study vasomotion at baseline and after exercise, hyperthermia and foot lowering within 3 groups of patients: diabetic without peripheral neuropathy, diabetic with subclinical peripheral neuropathy and diabetic with peripheral neuropathy and one group of sex- age- and body mass index-matched healthy control subjects.

All the subjects will benefit from a clinical, anthropometric, level of physical activity and biological evaluations. Type 2 diabetes participants will benefit from neuropathy evaluation. In addition, cutaneous microcirculation (perfusion and vasomotion) by means of Laser Doppler Flowmetry and Laser Speckle Imaging will be recorded at rest and after different stimuli (exercise, hyperthermia and foot lowering).

DETAILED DESCRIPTION:
All the subjects will benefit from a:

* clinical: diabetes duration, treatments
* anthropometric: weight, height, BMI
* level of physical activity by means of the International Physical Activity Questionary, pedometers and the 6 minutes walking test
* biological evaluations: glycemia, HbA1C, lipids, high sensitive C-reactive protein, fibrinogen, 25(OH)D, creatinine, albumine Type 2 diabetes participants will benefit from neuropathy evaluation: sensory tests by means of Semmes-Weinstein monofilament and of Nerve Check, amplitude and velocity sural nerve and neuropathic symptom score (NSS) In addition, cutaneous microcirculation (perfusion and vasomotion) by means of Laser Doppler Flowmetry and Laser Speckle Imaging will be recorded at rest and after different stimuli (exercise, hyperthermia and foot lowering).

ELIGIBILITY:
Inclusion Criteria:

* For diabetic patients, HbA1C >6.5 and diabetes duration >5years
* For healthy control no diabetes mellitus, no cardiovascular or renal pathology

Exclusion Criteria:

* nondiabetic neuropathy
* on medication known to affect microcirculation
* presence of active foot ulcer or wound healing history <3months
* inability to walk 6 minutes
* alcohol consumption of more than 3 units per day

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in average spectral amplitude of the entire frequency range between baseline and after stimulus | Cutaneous blood flow will be recorded during 20 minutes at rest, 10 minutes after foot lowering, 15 minutes after exercise and 20 minutes during hyperthermia
  Spectral analysis by wavelet analysis

CONTACTS AND LOCATIONS:
Overall Officials: Eric Benamo, MD, Principal Investigator — Centre Hospitalier Avignon
Locations (1):
- Centre Hospitalier Henri Duffaut, Avignon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynes C, Beaume JB, Latil-Plat F, Ennaifer H, Rocher L, Antoine-Jonville S, Benamo E, Knapp Y, Vinet A. Concomitant Peripheral Neuropathy and Type 2 Diabetes Impairs Postexercise Cutaneous Perfusion and Flowmotion. J Clin Endocrinol Metab. 2021 Sep 27;106(10):e3979-e3989. doi: 10.1210/clinem/dgab414. PMID 34111245